CLINICAL TRIAL: NCT07165171
Title: Glycemy After Periodontal Treatment in Patients With Type 2 Diabetes: a Randomized Controlled Trial Comparing Innovative Versus Standard Periodontal Follow-up
Brief Title: Periodontal Follow-up and Glycemy in Patients With Type 2 Diabetes
Acronym: GlyCoSup
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL23_0377; 2024-A01407-40 (Other: ID-RCB)
Record Dates: First submitted 2025-08-13; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Disease
Keywords: periodontal disease; Glycemy; Diabetes type 2; Follow-up
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Experimental comparative study to evaluate the effectiveness of a new strategy for monitoring type 2 diabetic patients who have been treated for periodontitis:
  - randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: SuP innovant (sending Short Message Service - SMS) (Experimental): For the Experimental Group: Innovative periodontal monitoring (SuP), consisting of:
  * visits every 3 months during 24 months with reinforcement of HBD advice and professional instrumentation - supra- and subgingival debridement if necessary. (common to the control group)
  * sending of different types of SMS: different types of SMS messages will be sent alternately.
  The SMS messages are intended for patients in the experimental group. The proposed approach aims to maintain contact with the patient at home and strengthen their commitment to a good oral hygiene routine over the long term. Text messages will be sent via the French CURECALL platform.
  The various text messages will be scheduled from the beginning of the periodontal follow-up.
  Interventions: Procedure: Innovative periodontal monitoring (SuP innovative)
- Control group: SuP standard (No Intervention): For the Control Group: Standard periodontal follow-up (SuP), consisting of: visits every 3 months with reinforcement of HBD advice and professional instrumentation - supra- and subgingival debridement if necessary (common to the experimental group).

INTERVENTIONS:
Procedure: Innovative periodontal monitoring (SuP innovative) — Different types of SMS messages will be sent alternately.
  * Type 1 SMS: SMS providing targeted medical information specifically for diabetic patients.
  * Type 2 SMS: Interactive SMS text messages written in the form of questions.
  * Type 3 SMS: Before each scheduled periodontal follow-up visit (every 3 months), a reminder SMS will be sent with the date, time, and location of the appointment.
  The SMS messages are intended for patients in the experimental group. Over these 24 months, the following are planned per patient:
  * 1 Type 1 SMS/week (medical advice or information);
  * 1 Type 2 SMS/month (interactive with suggested answers);
  * 1 Type 3 SMS every 3 months (appointment reminder): 1 per visit. The various text messages will be scheduled from the beginning of the periodontal follow-up.
  Other Names: Innovative periodontal monitoring (SuP innovative
  Arms: Intervention group: SuP innovant (sending Short Message Service - SMS)

SUMMARY:
Diabetes is a disease in which the majority of these patients have type 2 diabetes, linked to poor use of insulin by the body.

Periodontitis is a chronic disease characterized by an immuno-inflammatory reaction with local production of inflammatory mediators (IL6, TNF-alpha, etc.) and contributes to the increase in the systemic inflammatory load with increased levels of C-reactive protein.

Periodontitis is frequently found in diabetic patients; it is considered a complication of diabetes. Poor glycemic control in diabetes is associated with poor periodontal health, while periodontal infection is associated with dysglycemia and increased insulin resistance.

Periodontal treatment has been shown to reduce HbA1C levels and thus the risk of complications in diabetic patients.

The main objective is to evaluate the impact of innovative periodontal monitoring (with reminder systems and reinforcement of advice by SMS) versus standard periodontal monitoring on the glycemic control of diabetic patients treated for periodontitis, 2 years after the start of periodontal monitoring.

DETAILED DESCRIPTION:
Diabetes is a disease in which the majority of these patients have type 2 diabetes, linked to poor use of insulin by the body.

Periodontitis is a chronic disease characterized by an immuno-inflammatory reaction with local production of inflammatory mediators (IL6, TNF-alpha, etc.) and contributes to the increase in the systemic inflammatory load with increased levels of C-reactive protein.

Periodontitis is frequently found in diabetic patients; it is considered a complication of diabetes. Poor glycemic control in diabetes is associated with poor periodontal health, while periodontal infection is associated with dysglycemia and increased insulin resistance.

Periodontal treatment has been shown to reduce HbA1C levels and thus the risk of complications in diabetic patients.

However, periodontitis is a recurring disease; The implementation of periodontal monitoring (SuP) is essential throughout life after periodontal treatment, in order to prevent relapses. This monitoring, which must be carried out for life, includes the reassessment of periodontal criteria, professional instrumentation and oral hygiene (HBD) advice.

Visits every 3 months are generally recommended at the beginning, in order to regularly reinforce HBD advice. However, adherence to the SuP is difficult to obtain in the long term. In orthodontic patients, the use of reminder systems (SMS, emails, mobile applications, etc.) has a positive effect on HBD and periodontal criteria and would improve the rate of attendance at appointments in the medium term (3-12 months). A reminder and reinforcement system for HBD advice could therefore be integrated into the SuP in order to improve HBD and longer-term adherence in diabetic patients.

The main objective is to evaluate the impact of innovative periodontal monitoring (with reminder systems and reinforcement of advice by SMS) versus standard periodontal monitoring on the glycemic control of diabetic patients treated for periodontitis, 2 years after the start of periodontal monitoring.

This is a comparative experimental study to evaluate the effectiveness of a new monitoring strategy for type 2 diabetic patients who have been treated for periodontitis, a randomized controlled trial including an implementation study using a mixed methods approach (quantitative and qualitative).

The research will take place in 7 hospitals (Lille, Lyon, Nantes, Paris, Rennes, Strasbourg, Toulouse) and 7 privates dental centers in France.

Two types of care are proposed after periodontal treatment (all patients included will have previously benefited from standard periodontal treatment in the different centers).

The two groups compared will be:

* For the Experimental Group: Innovative periodontal monitoring.
* For the Control Group: Standard periodontal follow-up.

The primary endpoint is the HbA1c level (expressed in %) at 2 years after the date of randomization. The HbA1c level at 2 years will be collected by performing a routine dosage, in the patient's usual laboratory.

The target population of the GlyCoSuP project concerns adults with type 2 diabetes who have been treated for periodontitis.

After increasing by 10% to take into account those lost to follow-up, the total number of patients to be included will be 516 (258 patients per arm).

The duration of the inclusion period will be 24 months and the participation for each subject will be 24 months. In total, the total duration of the study will be 48 months.

ELIGIBILITY:
Inclusion Criteria:

* -- Adult aged 18 years or older;
* Presenting with type 2 diabetes (under ALD), balanced or not, for 6 months or more;
* Having been treated in the previous 6 months for periodontitis (stages 1 to 4 according to the new classification of periodontal and peri-implant diseases EFP-AAP 2018) in one of the participating centers and presenting a clinical situation allowing the transition to the periodontal follow-up phase (; (absence or limited number of sites presenting clinical signs of persistent periodontal inflammation)
* Presenting more than 6 teeth;
* Possessing a smartphone or tablet with internet access;
* Affiliated to social security;
* Patient able to read, write and understand French
* Having signed a consent to participate in the study.

Exclusion Criteria:

* Patient presenting uncontrolled systemic diseases and diagnosed for less than 6 months or presenting a major aggravation of a systemic pathology according to the judgment of the investigator.
* Pregnant or breastfeeding women;
* Persons deprived of liberty by a judicial or administrative decision;
* Adults subject to a legal protection measure (guardianship, curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c level (expressed as a %) | At 2 years after the date of randomization.
  The HbA1c level will be collected by routine testing in the patient's usual laboratory.
  This endpoint will be collected without knowing the patient's group. To limit missing data, a letter will be sent to the healthcare professional responsible for the patient's diabetes management (of the two groups) at the time of inclusion. If necessary, their physician may be contacted to retrieve this data, with the patient's consent.
  During the previous visit, the patient will be reminded to bring their test results for the next visit. This will also be noted in the appointment reminder text message.

SECONDARY OUTCOMES:
Periodontal criteria: - average probing depth (mm), | At inclusion and then every 3 months up to 24 months post-randomization.
  The periodontal probe used will be identical for all centers (purchase included in the study-funded budget): a manual periodontal probe with constant pressure, thus reinforcing standardization of practices.
  Collected by the investigator at inclusion and then every 3 months up to 24 months post-randomization.
Periodontal criteria: - bleeding index on probing (%), | At inclusion then every 3 months until up to 24 months post-randomization.
  The periodontal probe used will be identical for all centers (purchase included in the study-funded budget): a manual periodontal probe with constant pressure, thus reinforcing standardization of practices.
Periodontal criteria: - average clinical attachment level (mm), | At inclusion and then every 3 months up to 24 months post-randomization.
  The periodontal probe used will be identical for all centers (purchase included in the study-funded budget): a manual periodontal probe with constant pressure, thus reinforcing standardization of practices.
Periodontal criteria: - number of sites with a probing depth strictly greater than or equal to 4 mm (but with bleeding on probing), | at inclusion and then every 3 months up to 24 months post-randomization.
  The periodontal probe used will be identical for all centers (purchase included in the study-funded budget): a manual periodontal probe with constant pressure, thus reinforcing standardization of practices.
Periodontal criteria: - number of tooth loss, | at inclusion and then every 3 months up to 24 months post-randomization.
  The periodontal probe used will be identical for all centers (purchase included in the study-funded budget): a manual periodontal probe with constant pressure, thus reinforcing standardization of practices.
Periodontal criteria: - number of sites re-instrumented by debridement/root planing | at inclusion and then every 3 months up to 24 months post-randomization.
  The periodontal probe used will be identical for all centers (purchase included in the study-funded budget): a manual periodontal probe with constant pressure, thus reinforcing standardization of practices.
Diabetic Pathology Criteria: - HbA1c level (%), | At inclusion then every 3 months until 24 months post-randomization.
  HbA1c level (%): data collected from routine laboratory tests performed as part of diabetes management, in accordance with the recommendations of the French National Authority for Health (HAS), As a last resort, the physician may be contacted with the patient's consent to ensure that there have been no changes to the prescription since the last visit.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Hôpital Charles Foix, Ivry-sur-Seine
  - Centre Hospitalo-Universitaire de Lille, Lille
  - Hospices Civils de Lyon, Centre de Soins Dentaires., Lyon
  - Centre Hospitalo-Universitaire de Nantes, Nantes
  - Centre Hospitalo-Universitaire de Rennes, Rennes
  - Cabinet libéral, Saint-Victor-de-Cessieu
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Centre Hospitalo-Universitaire de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No